CLINICAL TRIAL: NCT04805112
Title: Acceptability, Feasibility and Impact of Oral HIV Self-testing for Partner Testing Among Kenyan Adolescent Girls Aged 15-19 Years: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Impact Research & Development Organization (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 848410
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV self-testing; partner testing; couples testing; transactional sex; young women; adolescent girls; female sex workers
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be recruited through the DREAMS (Determined, Resilient, Empowered, AIDS-Free, Mentored, Safe) program being implemented in Siaya County, western Kenya, as well as other community groups and venues, by the host institution (Impact Research and Development Organization, IRDO). Participants will be randomized in a 1:1 ratio to either an intervention group (receive multiple oral HIV self-test kits) or control (receive referral vouchers for clinic based testing). About 300 women will be recruited to patriciate in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Provision of multiple self-tests (Experimental): Participants randomized to the intervention group will be given 2-3 HIV oral self-tests to offer to their sexual partner(s). The participant will be instructed to encourage their partner to test himself alone [partner testing] or with the participant [couple testing]; the partner will also be given a card with information on testing and a list of facilities where he can go for confirmatory testing. All participants will be encouraged to call a study helpline/hotline in the event of any adverse events that they or their sexual partners experience or if they need further instructions or information
  Interventions: Behavioral: Provision of multiple self-tests
- Referral vouchers for clinic testing (No Intervention): Participants randomized to the control group will be given multiple referral coupons for HIV testing at pre-selected HIV testing services (HTS) sites. The participant will be instructed to give the coupon to their sexual partner(s) and encourage him to go for HIV testing at pre-selected HTS sites, either alone [partner testing] or together with the participant [couple testing]. The coupon will also have information on testing and a list of facilities where he can go for HTS. All participants will be encouraged to call a study helpline/hotline in the event of any adverse events that they or their sexual partners experience or if they need further instructions or information

INTERVENTIONS:
Behavioral: Provision of multiple self-tests — Participants will be given multiple Oraquick Advance HIV-1/2 test kits to distribute to their sexual partners for partner testing or couple testing. Phone interviews will be conducted with the participants to assess whether they provided a HIV self-test to their partner, if the test was used, how it was used (partner testing or couple testing), if the partner disclosed his results, the partner's reaction to the results, and if the partner went for confirmatory testing
  Arms: Provision of multiple self-tests

SUMMARY:
This randomized controlled trial will assess the feasibility, acceptability and impact of the provision of multiple oral-fluid based HIV self-test kits to HIV-negative adolescents aged 15-19 years to promote HIV testing among their sexual partners and couples testing.

DETAILED DESCRIPTION:
This study will recruit HIV-negative adolescents girls (AG) aged 15-19 years in Siaya County, western Kenya. The study will evaluate the impact of the provision of oral HIV self-testing on uptake of testing among partners of adolescent girls. We will randomize about 300 sexually active AG to either an intervention group that receives multiple oral self-test kits that they can choose to offer to their sexual partner(s) or to a control group that will be given multiple referral coupons that their partners can use for HIV testing at pre-selected HIV testing services (HTS) sites. We will collect data on whether the kits were offered, to whom they were offered, if they were accepted, if they were used and with what results, if known, and if the partners who obtained HIV-positive results sought confirmatory testing. We will also conduct in-depth interviews with a sub-set adolescents to explore their experiences in offering HIV self-testing to their male partners.

This study has 4 specific aims: i) determine whether adolescent girls can safely offer oral HIV self-tests to their partners; ii) assess whether oral self-testing improves uptake of HIV testing among partners of adolescent girls; iii) document adverse events associated with offering oral self-testing to sexual partners of adolescent girls; and iv) qualitatively explore the experiences of adolescent girls when offering self-test kits to their partners.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 15-19 years
* HIV-negative (willing to self-test onsite in the presence of the Research Assistant who is also a trained HIV counselor)
* Has at least one current sexual partner she expects to meet at least twice in the next 3 months (not necessarily to have sex); this will provide opportunity for the participant to suggest/offer testing.
* Resides in Siaya County and does not intend to relocate within 6 months from enrollment, to allow follow up to be completed and to conduct IDI with those selected.
* Willing to be randomized into the partner self-testing or HTS referral groups.
* Reporting no incident of sexual, physical, emotional, or economic abuse in the last 12 months from the partner she intends to offer (Appendix 4) or refer for testing (Appendix 3) in the next 3 months and does not believe the partner will abuse her if she offers the self-test kits or HTS referral coupon.
* Has a male partner who has not tested for 6 months or whose HIV status is unknown to her.
* Agrees to give consent to participate in the study.

Exclusion Criteria:

* Male
* HIV-positive
* Not willing to self-test onsite under in the presence of the Research Assistant
* Aged <15 years or >19 years
* Does not have a current sexual partner or does not expect to meet the partner at least twice in the next 3 months
* Does not reside in Siaya County or intends to relocate within the next 6 months
* Not interested in obtaining HIV self-tests or HTS referral coupon for purposes of suggesting testing to their sexual partners
* Reporting an incidence of sexual, physical, emotional or economic abuse in the last 12 months from the partner she would have offered self-test kit or referred for testing, or believes the partner may subject her to sexual, physical, emotional, or economic abuse if she offered them self-test kit or HTS coupon.
* Has a male partner who tested within the last 6 months.
* Does not give consent to participate in the study

Ages: 15 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 349 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
uptake of partner HIV testing | 3 months
  proportion of partners that complete HIV testing

SECONDARY OUTCOMES:
Introduce testing | 3 months
  proportion of participants who introduce testing to their partners
Partner accept testing | 3 months
  proportion of partners who were offered HIVST or referral coupon and accepted
Partner testing | 3 months
  proportion of participants who report their partner tested alone
Couples testing | 3 months
  proportion of participants who report testing with their partner
Positive partner | 3 months
  proportion of participants who report their partner test result was positive
linked to care | 3 months
  Proportion of participants who report their partners was linked to care
Intimate partner violence | 3 months
  proportion of participants in each study group who report intimate partner violence related to HIV testing
Confirmatory testing for positive HIV self-test | 3 months
  proportion of participants in the intervention group who report their partner tested positive and went for confirmatory testing

CONTACTS AND LOCATIONS:
Overall Officials: Kawango Agot, PhD, Principal Investigator — Impact Organization & Research Development; Harsha Thirumurthy, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Impact Research & Development Organization, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: No